CLINICAL TRIAL: NCT05569811
Title: A Phase 2 Trial of neoadjuVAnt muLti-agENT Chemotherapy or Patritumab Deruxtecan (HER3-DXd; U3-1402) With or Without endocrINE Therapy for High-risk HR+/HER2- Breast Cancer - VALENTINE Trial
Brief Title: NeoadjuVAnt muLti-agENT Chemotherapy or Patritumab Deruxtecan With or Without endocrINE Therapy for High-risk HR+/HER2- Breast Cancer - VALENTINE Trial
Acronym: VALENTINE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-2103; 2022-001181-36 (EudraCT Number)
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — patritumab deruxtecan; Drug Therapy; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHEMOTHERAPY (Active Comparator)
  Interventions: Drug: Chemotherapy
- HER3-DXd + Endocrine therapy (ET) (Experimental)
  Interventions: Drug: Patritumab deruxtecan; Drug: Letrozole
- HER3-DXd (Experimental)
  Interventions: Drug: Patritumab deruxtecan

INTERVENTIONS:
Drug: Patritumab deruxtecan — HER3-DXd will be administered as Lyo-DP, a sterile lyophilized powder in a dose of 5.6 mg/kg
  Arms: HER3-DXd; HER3-DXd + Endocrine therapy (ET)
Drug: Chemotherapy — Anthracycline/taxane-based neoadjuvant regimen recommended by the NCCN or local guidelines. i.e. EC or AC (epirubicin 90 mg/m2 or doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 every 14 or 21 days) followed by weekly paclitaxel 80mg/m2 during 12 weeks
  Arms: CHEMOTHERAPY
Drug: Letrozole — Letrozole and LHRH will be used following SmPC specifications, according to standard therapy and clinical studies
  Arms: HER3-DXd + Endocrine therapy (ET)

SUMMARY:
VALENTINE is a parallel, non-comparative, three-arm, randomized 1:2:2 open-label, multicenter, exploratory study in women or men with primary operable HR+/HER2-negative breast cancer with ki67 ≥ 20% and/or high genomic risk (defined by gene signature) aiming at evaluating the clinical benefit and biological effects of HER3-DXd with/without letrozole as a neoadjuvant treatment regimen.

The primary aim is to evaluate the ability of each treatment strategy to achieve a pCR at surgery. This study is exploratory and no formal comparison between treatment arms is intended. The inclusion of a chemotherapy treatment arm serves as an internal response control instead of using historical data as comparators. In addition, the chemotherapy control arm is the standard of care appropriate treatment in these patients, to include this arm will ensure the recruitment of the target patient population (patients should have indication for neoadjuvant chemotherapy) and allowing comparison of secondary endpoint such as safety and/or HrQoL.

ELIGIBILITY:
Main inclusion criteria

1. Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast untreated and recently diagnosed
2. ER-positive and/or PgR-positive and HER2-negative tumor
3. Ki67% ≥ 20% locally assessed and/or high genomic risk (defined by gene signature):
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
5. Breast cancer eligible for primary surgery.
6. Availability of pre-treatment tumor tissue sample of FFPE tumor block from primary tumor for biomarker analysis.
7. Participants must be deemed eligible for neoadjuvant chemotherapy
8. Participants must be deemed eligible for surgery.
9. Adequate hematologic and end-organ function, defined by the following laboratory results
10. Baseline LVEF ≥ 50% measured by echocardiography (ECHO) or Multiple Gate Acquisition (MUGA) scan

Main exclusion criteria

1. Metastatic (Stage IV) breast cancer.
2. Bilateral invasive breast cancer.
3. Any treatment, local or systemic, including prior chemotherapy, ET, targeted therapy, and/or radiation therapy for the currently diagnosed BC prior to enrollment.
4. Patients in whom a primary tumor excisional biopsy was performed.
5. Prior treatment with a HER3 antibody, topoisomerase I inhibitor, with an ADC which consists of an exatecan derivative that is a topoisomerase I inhibitor (e.g., DS-8201) and with a govitecan derivative (e.g., IMMU-132).
6. Patient has active cardiac disease or a history of cardiac dysfunction.
7. Medical history of clinically significant lung diseases (e.g., interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) or who are suspected to have these diseases by imaging at screening period.
8. Patients with a history of any malignancy are ineligible except specific cases
9. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary or metabolic disease; wound healing disorders; ulcers; bone fractures, psychiatric illness/social situations, geographical factors, substance abuse) or other factors which in the Investigator's opinion makes it undesirable for the subject to participate in the study or which would jeopardize compliance with the protocol
10. Concurrent, serious, uncontrolled infections or current known infection with HIV or active hepatitis B and/or hepatitis C.
11. History of significant co-morbidities that, in the judgment of the investigator, may interfere with the conduction of the study, the evaluation of response, or with ICF.
12. Known hypersensitivity to either the drug substance components (including an antibody, a drug-linker, or a topoisomerase I inhibitor) or inactive ingredients in the drug product or history of severe hypersensitivity reactions to other monoclonal antibodies.
13. History of exposure to cumulative anthracycline doses greater than follows: a. Adriamycin > 100 mg/m2; Epirubicin > 180 mg/m2; Mitoxantrone > 40 mg/m2; Idarubicin > 22.5 mg/m2. If another anthracycline or more than one anthracycline has been used, the cumulative dose must not exceed the equivalent of 100 mg/m2 of adriamycin.
14. Any history of interstitial lung disease (ILD) (including pulmonary fibrosis or radiation pneumonitis), has current ILD, or is suspected to have such disease by imaging during screening.
15. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorders with potential pulmonary involvement (i.e. rheumatoid arthritis, Sjögren's syndrome, sarcoidosis etc.), or prior pneumonectomy.
16. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, grade ≤1 or baseline. Subjects with chronic grade 2 toxicities may be eligible per the discretion of the Investigator.
17. Non-eligible for taxanes therapy. Previous sensory neuropathy > grade 1, according to NCI-CTCAE criteria, due to any reason.
18. Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to Cycle 1 Day 1. Subjects who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study.
19. Evidence of any leptomeningeal disease.
20. Has clinically significant corneal disease.
21. Female subject who is pregnant or breastfeeding or intends to become pregnant during the study.
22. Subjects who are currently receiving chloroquine or hydroxychloroquine. A washout period of > 14 days is required prior to randomization or Cycle 1 Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pCRBL (ypT0/is ypN0) at surgery | before treatment and surgery
  complete absence of invasive carcinoma in the breast and axillary lymph nodes on histological examination.

SECONDARY OUTCOMES:
Rate of Residual cancer burden (RCB) category status (0, I, II, III) | before treatment and surgery
  assessed by a local pathologist at surgery according to the MD Anderson Cancer Center recommendations.
pCRB (pathological complete response in the breast) | before treatment and surgery
  defined as the complete absence of invasive carcinoma in the breast on histological examination after treatment, irrespective of in situ carcinoma in the breast.
Tumor overall objective response rate (ORR) | before treatment and pre-surgery
  defined as the proportion of subjects with a Partial Responses (PR) or a Complete Responses (CR) according to RECIST v1.1 as per Investigator's assessments by breast MRI
iDFS rate | 3 years follow-up and 5 years follow-up
  iDFS defined as the time from randomization to any of the following events:
  * Ipsilateral invasive breast tumor recurrence (IIBTR): invasive breast cancer involving the same breast parenchyma as the original primary.
  * Regional invasive breast cancer recurrence: Invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast.
  * Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer.
  * Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
  * Contralateral invasive breast cancer.
  * Second primary non-breast invasive cancer.
  * Progression during neoadjuvant treatment.
CelTIL score changes | from baseline to C2D1
  CelTIL score (CelTIL = = -0.8 × tumor cellularity (in %) + 1.3 × TILs (in %)
HER3 receptor expression and ERBB3 mRNA expression level | from baseline to C2D1
  HER3 receptor expression levels by IHC and ERBB3 mRNA expression level by gene expression.
Proliferation | from baseline to C2D1
  changes in ki67 IHC
Quality of Life assessed by EORTC-BR45 changes | from baseline until 30 days after the surgery visit
  European Organization for Research and Treatment of Cancer's (EORTC) core quality for assessing quality of life in breast cancer patients (EORTC-BR45). QLQ-BR45 is used to measure HRQoL within the preceding 7 days or 28 days depending on the items. The EORTC QLQ-BR45 is a questionnaire consisting of 45 items where each item is scored using a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much).
Quality of Life assessed by EORTC QLQ-C30 changes | from baseline until 30 days after the surgery visit
  European Organization for Research and Treatment of Cancer's (EORTC) core quality of life questionnaire (EORTC QLQ-C30, version 3.0). EORTC QLQ-C30 is used to measure QoL within the preceding 7 days. The EORTC QLQ-C30 is a questionnaire consisting of 30 items where each item is scored using a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much).
Number of Participants with Adverse events (safety) | from randomization/enrollment to end of safety follow up assessed up to approximately 30 days after the surgery visit
  Type, incidence, severity (as graded by the NCI CTCAE v. 5.0), seriousness and attribution to the study medications of TEAEs, AESI and any laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (25):
- Spain (25):
  - ICO Badalona, Badalona, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, La Coruña
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General de Catalunya, Barcelona
  - Hospital Universitari Vall d' Hebrón, Barcelona
  - Hospital de Basurto, Bilbao
  - Complejo Hospitalario San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - H.Univ. Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - HAU de Manresa, Manresa
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Sant Joan de Reus, Reus
  - HU Parc Tauli, Sabadell
  - Comp. Hosp.Univ. Santiago (Chus), Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - H La Fe, Valencia
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.gruposolti.org/